CLINICAL TRIAL: NCT03768011
Title: A Subjective Observational Study of Patients Using Transdermal Cream Medication And/Or Transdermal Patches With Or Without Oral Non-Narcotic Medications to Help Reduce or Eliminate Use of Opiates
Brief Title: Subjective Observational Study of Patients Using Transdermal Cream Medication And/Or Transdermal Patches With Or Without Oral Non-Narcotic Medications
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Data Collection Analysis Business Management (Other)
Responsible Party: Sponsor
Other Study IDs: PAS1466
Record Dates: First submitted 2018-12-01; First posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Pain, Chronic; Pain, Joint; Pain Syndrome
MeSH Terms: conditions — Chronic Pain; Arthralgia; Somatoform Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: transdermal cream and or patch — transdermal cream and/or transdermal patch(s) with or without oral medication

SUMMARY:
purpose of this study is to evaluate the level of pain perceived by patients using a transdermal cream and/or transdermal patch with or without an oral medication as a pain management solution.

DETAILED DESCRIPTION:
The purpose of this minimal risk, observational study is to observe and document patients' perspective on how the combination of transdermal cream and/or transdermal patch(s) with or without oral medication can help reduce or eliminate the use of opiate(s).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be diagnosed with an ICD10 code indicative of chronic pain
* Participants must be starting a new regimen of topical therapy with or without non-narcotic oral medication that has been deemed medically necessary and is independent of the study
* Participants must be expecting to receive therapy for at least 12 weeks
* Participants must be between 18 and 64 years of age
* Participants must be able to provide sound verbal informed consent

Exclusion Criteria:

* Participants must not be a beneficiary of government funded healthcare program (i.e. Medicare, Medicaid, etc.)
* Participants must not have a diagnosis of cancer within the past 5 years
* Participants who have chronic pain conditions not expected to respond to topical pain medication such as deep abdominal pain, or from conditions such as cancer

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: a patient with joint pain, extremity pain, lumbar, thoracic and/or cervical pain, as part of the PI routine care or follows medical necessity and prescribes a combination topical cream and/or patch with or without non-narcotic oral medication independent of the study
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Patients' perspective through a patient led Survey of Health and quality of life via patient reported outcome measures using Visual analogue scale given at Baseline and follow up. Measuring pain from 0 no pain to 10 highest pain level. | 36 months
  Collecting and analyzing quantitative and qualitative data to draw generalized outcome measures, on real world data.Data from the subject surveys will analyze and measure the effectiveness through a subjective observation via patients' perspective survey on transdermal cream and/or transdermal patches with or without oral non-narcotic medication and if it helped with the reduction or elimination of opiate(s).

SECONDARY OUTCOMES:
Visual Analogue scales | 36 months
  By utilizing the Visual analogue scale from the patients' perspective will generate real world data

CONTACTS AND LOCATIONS:
Locations (1):
- DCABM, Land O' Lakes, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided